CLINICAL TRIAL: NCT04216173
Title: Acupuncture for Headache Post-Traumatic Brain Injury: A Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Permanent suspension of all study activities due to COVID-19 and subsequent loss of funding.
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Mark Sodders, Post Doctoral Scholar, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00008281; KL2TR002317-03S1 (NIH)
Record Dates: First submitted 2019-12-14; First posted 2020-01-02 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Post-Traumatic Headache; Traumatic Brain Injury
Keywords: Acupuncture; Post-traumatic headache; Traumatic brain injury
MeSH Terms: conditions — Post-Traumatic Headache; Brain Injuries, Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture weekly for 12 consecutive weeks. Acupuncture protocol consists of both scalp and body acupuncture points.

SUMMARY:
This study evaluates and addresses challenges to implementing an acupuncture intervention for adults who have headaches after sustaining a moderate traumatic brain injury. Eligible participants will be recruited from Seattle and the surrounding areas to receive weekly acupuncture for 12 consecutive weeks. Participants will complete questionnaires to assess headache impact, depression, health-related quality of life, and cognitive function at the beginning of the study and every two weeks for the duration of the study. Participants will participate in structured interviews after the study for their views on the acceptability and tolerability of the study protocol.

ELIGIBILITY:
Inclusion Criteria

* Has a history of moderate traumatic brain injury (TBI) one to five years previously
* Currently under medical supervision for post-traumatic headache
* Have a score ≥ 3 on the Patient Health Questionnaire 2
* Have a raw summed score ≤ 6 on the PROMIS Cognitive Function Short Form v2.0 - Abilities 2a (part of PROMIS-29+2 Profile)
* Community-dwelling
* 18 years of age and older
* English Speaking
* Able to provide voluntarily consent

Exclusion Criteria

* History of multiple TBIs
* History of receiving acupuncture treatment in the past six months for the primary condition of headache
* An established diagnosis of PTSD
* Psychosis or agitation
* Other neurodegenerative disorders
* Other medical/surgical condition that precludes travel to participate in the intervention over the study duration
* Has an active skin lesion or acute trauma over or around the proposed acupuncture points
* History of trauma to the head that currently prevents the use of acupuncture points along the midline of the scalp
* Persons who are pregnant
* Unable to provide informed consent for the research as identified as answering more than two incorrect responses on the Six-item Screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Proportion of weekly acupuncture sessions completed over 12 consecutive weeks | 12 weeks
  Retention rate will be evaluated by the proportion of weekly acupuncture sessions completed per participant over the course of 12 consecutive weeks.
Proportion of survey questionnaires completed | Baseline
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 2 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 4 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 6 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 8 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 10 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Proportion of survey questionnaires completed | 12 weeks
  Respondent burden will be evaluated by the proportion of survey questionnaires completed.
Data completeness in survey questionnaires | Baseline
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 2 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 4 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 6 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 8 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 10 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Data completeness in survey questionnaires | 12 weeks
  Data completeness in survey questionnaires will be evaluated during data collection.
Participants' perceptions of feasibility of the study with structured interviews | After 12 weeks, or within two weeks of withdrawal from the study
  After 12 weeks in the study, participants will participate in structured interviews for their views on the acceptability and tolerability of the study protocol and acupuncture protocol, recommendations for recruitment and retention, and experiences during the intervention. Interviews with participants withdrawn from the study will be attempted within two weeks of the withdrawal.

SECONDARY OUTCOMES:
Headache Impact Test - 6 | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  A brief measure describing how a headache affects a participant's functional health and well-being. Score ranges from 36 to 78. Higher scores indicate worse outcomes.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  A measure of depression severity. Scores may range from zero to 27. Higher scores indicate worse outcomes.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of depression collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Higher scores indicate worse outcomes.
PROMIS Short Form v1.0 - Anxiety 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of anxiety, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Higher scores indicate worse outcomes.
PROMIS Short Form v2.0 - Physical Function 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of physical function, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Lower scores indicate worse outcomes.
PROMIS Short Form v1.0 - Pain Interference 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of pain interference, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Higher scores indicate worse outcomes.
PROMIS Short Form v1.0 - Fatigue 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of fatigue, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Higher scores indicate worse outcomes.
PROMIS Short Form v1.0 - Sleep Disturbance 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of sleep disturbance, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Higher scores indicate worse outcomes.
PROMIS Short Form v1.0 - Ability to Participate in Social Roles and Activities 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of one's ability to participate in social roles and other activities, collected as a part of the PROMIS-29 v2.1 profile. There are four questions, with a possible score of four to 20. Lower scores indicate worse outcomes.
PROMIS Pain Intensity Item (Global07) | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of pain intensity, collected as a part of the PROMIS-29 v2.1 profile. This is a single question, with a possible score of 0 to 10. Higher scores indicate worse outcomes.
PROMIS Short Form v2.0 - Cognitive Function 4a | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Participant reported measure of cognitive function. There are four questions, with a possible score of four to 20. Lower scores indicate worse outcomes.
Self-reported changes in medication dose | Baseline, 12 weeks
  Changes in medication

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Sodders, DOAM, Principal Investigator — University of Washington
Locations (1):
- Harborview Injury Prevention and Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No